CLINICAL TRIAL: NCT03948178
Title: Effects of Oral Levosimendan (ODM-109) on Respiratory Function in Patients With ALS: Open-Label Extension for Patients Completing Study 3119002
Brief Title: Effects of Oral Levosimendan on Respiratory Function in Patients With Amyotrophic Lateral Sclerosis (ALS): Open-Label Extension
Acronym: REFALS-ES
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This was an open label extension for patients completing the REFALS study (3119002; NCT03505021). Study 3119002 showed lack of efficacy of ODM109 so the sponsor decided to terminate this study
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3119003
Record Dates: First submitted 2019-05-07; First posted 2019-05-13 (Actual); Results first posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Simendan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Levosimendan (Experimental): Oral Levosimendan; Levosimendan 1mg capsules for oral administration, once to twice a day, continued as long as clinically beneficial. The total study duration is up to 3 years.
  Interventions: Drug: Levosimendan

INTERVENTIONS:
Drug: Levosimendan — Levosimendan 1 mg capsule for oral administration
  Other Names: ODM-109

SUMMARY:
This study provides an opportunity for subjects in the REFALS (3119002; NCT03505021) study to continue treatment with oral levosimendan. The study will also provide more information about long-term safety and effectiveness of oral levosimendan in patients with ALS.

This is an open-label study, so that all eligible subjects that complete the double-blind REFALS study (48-weeks of treatment) will have the opportunity to receive oral levosimendan treatment. The primary objective, in addition to continuing treatment for subjects enrolled in the REFALS study, is to evaluate long-term safety of oral levosimendan in ALS patients. Another important objective is to explore long-term effectiveness of oral levosimendan in the treatment of patients with ALS.

This study is open only to patients taking part in the REFALS study.

ELIGIBILITY:
Inclusion Criteria:

* Written or verbal informed consent (IC) for participation in the study
* Subjects who completed 48 weeks of treatment according to the REFALS study protocol
* Able to swallow study treatment capsules at the time of completing 48 weeks dosing in the REFALS study

Exclusion Criteria:

* Development (or significant worsening from baseline of the REFALS study) of serious cardiovascular disease (e.g.: myocardial infarction, heart failure, arrhythmia, stroke, or second or third degree atrioventricular (AV) block)
* Pulse/heart rate repeatedly >100 bpm after 5-minute rest at baseline. If the pulse/heart rate is >100 bpm in the first recording, then a second recording must be done after another 5 min rest to confirm pulse/heart rate >100 bpm
* Systolic blood pressure (SBP) <90 mmHg
* Severe renal impairment (creatinine clearance < 30ml/min or creatine >170 µmol/l at 48 week visit of the REFALS study, or on dialysis
* Severe hepatic impairment at the discretion of the investigator
* Women of reproductive age without a negative pregnancy test and without a commitment to using a highly effective method of contraception (e.g.: oral hormonal contraceptive associated with inhibition of ovulation, intrauterine devices and long acting progestin agent), if sexually active during the study, and for 1 month after the last dose of the study treatment. Women who are postmenopausal (1 year since last menstrual cycle), surgically sterilised or who have undergone a hysterectomy are considered not to be reproductive and can be included
* Subject judged to be actively suicidal by the investigator
* Any other clinical significant cardiovascular, gastrointestinal, hepatic, renal, neurological or psychiatric disorder or any other major concurrent illness that in the opinion of the investigator could interfere with the interpretation of the study results or constitute a health risk for the subject if he/she took part in the study

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2020-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève Nadeau, CSD, Study Director — Orion Corporation, Orion Pharma
Locations (79):
- United States (31):
  - Neuromuscular research Centre and Neuromuscular Clinic of Arizona, Phoenix, Arizona
  - University of California San Diego, La Jolla, California
  - University of California Irvine Medical Center, Orange, California
  - Hospital for Special Care, New Britain, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - The George Washington Medical Faculty Associates, Washington D.C., District of Columbia
  - Holy Cross Hospital Neuroscience Institute, Fort Lauderdale, Florida
  - University of Florida McKnight Brain Institute, Gainesville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of South Florida/USF Health, Tampa, Florida
  - Augusta University, Medical Centre, Augusta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Michigan Medicine University Hospital, Ann Arbor, Michigan
  - Health Partners Speciality Center, Saint Paul, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Neurology Associates, Lincoln, Nebraska
  - Hospital for Special Surgery, New York, New York
  - Columbia Presbyterian Hospital, New York, New York
  - Neurosciences Institute - Neurology Charlotte, Charlotte, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - The Ohio State University Wexner Medical center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Providence Brain and Spine Institute, Portland, Oregon
  - Alleghenay General hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Nerve and Muscle Centre of Texas, Houston, Texas
  - University of Utah Health-Imaging & Neurosciences Center in research Park, Salt Lake City, Utah
  - University of Washington Medical Center, Seattle, Washington
- Australia (5):
  - Brain and Mind Centre, Camperdown, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Calvary Health Care Bethlehem, Parkdale, Victoria
  - Perron Institute for Neurological and Translational Science, Nedlands, Western Australia
- Austria (3):
  - Medizinische Universitat Innsbruck, Innsbruck, Tyrol
  - Salzqammergut-klinikum Vocklabruck, Neurologie, Vöcklabruck, Upper Austria
  - Medizinische Universitat wein Universitatsklinik ffur Neurologie, Wein
- Belgium (3):
  - Algemeen Ziekenhuis St Lucas Gent, Ghent
  - Universitair Ziekenhuis Leuven, Leuven
  - Centre Hospitalier Regional de la Vitadelle, Liège
- Canada (7):
  - Alberta Health Services-Neuromuscular Clinic, Calgary, Alberta
  - University of Alberta, Division of Neurology, Edmonton, Alberta
  - Stan Cassidy Centre for Rehabilitation, Fredericton, New Brunswick
  - McMaster University Medical Centre, Hamilton, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
  - Centre Hospitalier Affilie Universitaire de Quebec, Québec, Quebec
- Finland (2):
  - Helsinki University Central Hospital, Neurology Outpatients Clinic, Helsinki
  - Turku University Hospital, Turku
- France (3):
  - Centre Hospitalier Universitaire de Limoges Service de Neurologie, Limoges
  - Hopital Gui de Chauliac Service de Neurologie, Montpellier
  - Hopital Pasteur Centre de reference des Malades Neuromusculaires et SLA, Nice
- Germany (7):
  - Charite Universitatmedizin Berlin- Campus Virchow-Klinikum, Berlin
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum Jena, Klinik fur Neurologie, Jena
  - Universitatsklinikum Munster, Institut fur Schalfmedizin und Neuromuskalaire Erkrankungen, Münster
  - Universitatsmedizin Rostock, Klinik und Poliklinik fuer Neurologie, Rostock
  - Universitatsklinikum Ulm, Poliklinik fur Neurologie, Ulm
  - Deutsche Klinik fur Daignostik, Wiesbaden
- Beaumont Hospital, Clinical Research Centre, Dublin, Ireland
- Italy (6):
  - Azienda Policlinico San Martino, Genova
  - ICS Maugeri Spa S UO Riabilitazione Nurologica, Milan
  - Azienda Ospedaliera Universitaria-maggiore della Carita di Novara, Novara
  - Azienda Ospedaliero Universitaria Pisana Ospedale Santa Chiara, Pisa
  - Policlinico Umberto I di Roma Clinica Neurologica, Rome
  - Azienda Ospedaliera Universitaria Citta della Salute e della Scienza di Torino, Torino
- Univeritair Medisch Centrum Utrech, Utrecht, Netherlands
- Spain (5):
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Hospital Universitario Reina Sofia Servicio Neurologia, Córdoba
  - Hospital San Rafael, Madrid
  - Hospital Universitario y Politecnico de La Fe, Valencia
- Sweden (3):
  - Karlstad Central Hospital Neurology and Rehabilitation, Karlstad
  - Karolinska University Horpital Huddinge Neurology Clinic, Stockholm
  - Norrlanda University Hospital Neuro-huvud-hals-centrum Vasterbotten, Umeå
- United Kingdom (2):
  - The Walton Centre NHs Foundation Trust, Neurology and Neurosurgery, Liverpool
  - Barts Health NHS Trust Royal London hospital, London

REFERENCES:
- [Derived] Cudkowicz M, Genge A, Maragakis N, Petri S, van den Berg L, Aho VV, Sarapohja T, Kuoppamaki M, Garratt C, Al-Chalabi A; REFALS investigators. Safety and efficacy of oral levosimendan in people with amyotrophic lateral sclerosis (the REFALS study): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet Neurol. 2021 Oct;20(10):821-831. doi: 10.1016/S1474-4422(21)00242-8. PMID 34536404

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with amyotrophic lateral sclerosis (ALS) who completed 48 weeks of treatment in the REFALS study (NCT03505021) were recruited
Pre-assignment Details: Male or female subjects with a diagnosis of probable or definite ALS having completed 48 weeks of treatment in the REFALS Study (NCT03505021) and able to swallow study treatment capsules at the time of completing 48 weeks of dosing in the REFALS study. Written or verbal informed consent obtained.
Period: Overall Study
Arm/Group | Levosimendan
Started | 227
Completed | 0
Not Completed | 227
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2
Not completed — Reason not known | 2
Not completed — Personal reason | 14
Not completed — Disease progression | 30
Not completed — Adverse Event | 12
Not completed — Sponsor terminated study | 164

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat (ITT) including all randomised subjects was used for the primary evaluation.
Arm/Group | Levosimendan
Number analyzed (Participants) | 227
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 160
  >=65 years | 67
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 224
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 218
  More than one race | 0
  Unknown or Not Reported | 9

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events Recording
Description: Adverse Events as subject counts and proportions (%) of subject per Adverse Event
Time Frame: From signing informed consent until 14-25 days after the last study treatment for all patients, an average of 23.5 weeks.
Population: Analysis is reported for the safety population which included all subjects receiving any study treatment. Treatment emergent AEs are defined as any event arising or worsening after the start of study treatment until 25 days after the individual subject's last study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Levosimendan
Number analyzed (Participants) | 227
Participants | 161

2. Primary Outcome: Pulse/Heart Rate Assessment
Description: Actual values and changes from baseline in supine pre-dose pulse/heart rate were summarised using descriptive statistics .
Time Frame: Change in pulse and heart rate(from ECG recording) from Baseline, week 2, week 4, week 6 (pulse rate only), Month 3, Month 6, end of study (subject's last visit, 2-48 weeks after study entry)
Population: Analysis was performed on the safety population which included all patients who had received at least one dose of study treatment. The change from baseline in pulse and heart rate was measured at week 2, week 4, week 6 (pulse rate only) Month 3, Month 6 and the individual subject 's last visit in the study. The number of subjects analysed at each timepoint differs from the total number of subjects that entered the study as some study subjects did not undergo the assessment at all timepoints.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Levosimendan
Number analyzed (Participants) | 224
beats per minute (bpm)
  Change in pulse rate at week 2: number analyzed (Participants) | 218
  Change in pulse rate at week 2 | 7.0 (8.8)
  Change in pulse rate at 4 weeks: number analyzed (Participants) | 180
  Change in pulse rate at 4 weeks | 10.0 (10.4)
  Change in pulse rate at week 6: number analyzed (Participants) | 196
  Change in pulse rate at week 6 | 8.5 (12.0)
  chnage in pulse rate at Month 3: number analyzed (Participants) | 121
  chnage in pulse rate at Month 3 | 10.4 (10.6)
  Change in pulse rate at month 6: number analyzed (Participants) | 57
  Change in pulse rate at month 6 | 12.8 (10.6)
  Change in pulse rate at end-of-study: number analyzed (Participants) | 173
  Change in pulse rate at end-of-study | 3.5 (12.6)
  Change in Heart rate at week 2: number analyzed (Participants) | 157
  Change in Heart rate at week 2 | 9.1 (10.1)
  Change in Heart rate at week 4: number analyzed (Participants) | 106
  Change in Heart rate at week 4 | 12.8 (9.4)
  Change in heart rate at Month 3: number analyzed (Participants) | 75
  Change in heart rate at Month 3 | 12.6 (9.3)
  Change in heart rate at month 6: number analyzed (Participants) | 40
  Change in heart rate at month 6 | 15.0 (9.9)
  Change in heart rate at end-of-study: number analyzed (Participants) | 109
  Change in heart rate at end-of-study | 5.3 (10.9)
  Baseline supine pulse rate | 75.8 (12.5)
  Baseline supine heart rate: number analyzed (Participants) | 193
  Baseline supine heart rate | 73.5 (12.0)

3. Primary Outcome: 12-lead Electrocardiogram Assessments
Description: Summarisation of any abnormal 12-lead ECG findings using descriptive statistics.
Time Frame: Baseline, week 2, week 4, month 3, month 6, end-of-study(subject's last visit, 2-48 weeks after study entry)
Population: Analysis of patients in the safety population defined as all patients who had received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Levosimendan
Number analyzed (Participants) | 227
Participants
  Baseline abnormal ECG | 69
  Week 2 abnormal ECG | 56
  Week 4 abnormal ECG | 43
  Month 3 abnormal ECG | 27
  Month 6 abnormal ECG | 11
  End-of study abnormal ECG | 36

4. Secondary Outcome: Disease Progression
Description: Count of study withdrawals due to disease progression
Time Frame: From Baseline through study completion(subject's last visit, 2-48 weeks after study entry)
Population: Number of study withdrawals due to disease progression were collected for all subjects entered into the study. The study sponsor terminated the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Levosimendan
Number analyzed (Participants) | 227
Participants
  Total withdrawal due to sponsor terminating the study | 164
  Number of withdrawals due to disease progression | 30

5. Secondary Outcome: Supine Slow Vital Capacity (SVC)
Description: Change from baseline in supine and sitting SVC (all devices) through to the end of the study, expressed as a % of predicted normal
Time Frame: The change from Baseline, week 2, week 4, month 3, month 6, end-of-study (subject's last visit, 2-48 weeks after study entry)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % of predicted normal
Arm/Group | Levosimendan
Number analyzed (Participants) | 185
% of predicted normal
  Change from baseline in supine SVC at week 2: number analyzed (Participants) | 133
  Change from baseline in supine SVC at week 2 | 1.5 (7.2)
  Change from baseline in supine SVC at week 4: number analyzed (Participants) | 89
  Change from baseline in supine SVC at week 4 | 0.8 (10.2)
  Change from baseline in supine SVC at month 3: number analyzed (Participants) | 62
  Change from baseline in supine SVC at month 3 | -3.5 (10.4)
  Change from baseline in supine SVC at month 6: number analyzed (Participants) | 30
  Change from baseline in supine SVC at month 6 | -5.3 (13.2)
  Change from baseline in supine SVC at the end of the study: number analyzed (Participants) | 57
  Change from baseline in supine SVC at the end of the study | -5.6 (17.4)
  Change from baseline in sitting SVC at week 2: number analyzed (Participants) | 139
  Change from baseline in sitting SVC at week 2 | 1.4 (6.6)
  Change from baseline in sitting SVC at week 4: number analyzed (Participants) | 91
  Change from baseline in sitting SVC at week 4 | 2.1 (9.8)
  Change from baseline in sitting SVC month 3: number analyzed (Participants) | 65
  Change from baseline in sitting SVC month 3 | -1.9 (11.9)
  Change from baseline in sitting SVC month 6: number analyzed (Participants) | 33
  Change from baseline in sitting SVC month 6 | -6.1 (12.4)
  Change from baseline in sitting SVC at the end of the study: number analyzed (Participants) | 77
  Change from baseline in sitting SVC at the end of the study | -7.3 (12.1)
  Baseline Supine SVC (% predicted normal | 54.4 (21.6)
  Baseline Sitting SVC (% predicted normal): number analyzed (Participants) | 176
  Baseline Sitting SVC (% predicted normal) | 61.4 (19.4)

6. Secondary Outcome: Revised ALS Functional Rating Scale (ALSFRS-R)
Description: ALSFRS-R scale contains 3 parameters related to respiratory function: Severity of dyspnea, occurrence of orthopnea (shortness of breath when in supine position i.e. lying flat), and the use of mechanical ventilation for respiratory in sufficiency. These 3 parameters are combined to create the respiratory domain with a score of 0-12(where 12 is normal function). Although individual items and patients vary, ALSFRS-R typically declines at a relatively constant rate over time. Plotted over time the slope of the line obtained indicates the speed of progression and thus an effective treatment might be expected ro reduce the slope of decline.
Time Frame: Change from Baseline in respiratory function of ALSFRS-R at study completion (subject's last visit, 2-48 weeks after study entry)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Levosimendan
Number analyzed (Participants) | 226
Score on a scale
  Change from baseline in respiratory function ALSFR-S at end of study: number analyzed (Participants) | 192
  Change from baseline in respiratory function ALSFR-S at end of study | -1.2 (2.3)
  Baseline respiratory ALSFRS-R | 9.4 (3.0)

7. Secondary Outcome: Need for Respiratory Support Device
Description: Time to respiratory device support (non invasive) or death
Time Frame: Time to event at study completion (subject's last visit, 2-48 weeks after study entry)
Population: Analyses were performed in the safety population in which all subjects received at least one dose of study treatment
Measure: Mean (Standard Error); unit: days
Arm/Group | Levosimendan
Number analyzed (Participants) | 227
days | 259.5 (10.46)

8. Secondary Outcome: Borg Category Ratio 10 Scale (CR 10)
Description: Patients rated their perception of the severity of their dyspnea using the Borg Category Ration 10 scale (CR 10). The scale ranges from 0(no dysponea) to 10 (maximal dyspnea). each category is numbered and most but not all have verbal cues. At each assessment the patient scored the category they felt best described their symptoms. The analysis measured change from baseline to the end of the study in both a supine and sitting position where a negative score indicates improvement and a positive score reflects worsening.
Time Frame: Baseline through study completion (week 2, week 4, month 3, month 6, end of study (subject's last visit, 2-48 weeks after study entry)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levosimendan
Number analyzed (Participants) | 203
units on a scale
  Baseline in Borg score Supine position | 2.52 (2.62)
  Change from baseline in Borg score supine at week 2 | 0.15 (2.16)
  chenge from baseline in Borg score week 4 | 0.40 (2.21)
  Change from baseline in Borg score supine at month 3 | 0.54 (2.05)
  Change from baseline in Borg score supine at month 6 | 1.61 (2.07)
  Change from baseline in Borg score supine at end of study | 1.58 (2.78)
  Baseline Borg score sitting: number analyzed (Participants) | 202
  Baseline Borg score sitting | 2.19 (2.33)
  Change from baseline in Borg score sitting at week 2 | 0.01 (1.71)
  Change from baseline in Borg score sitting at week 4: number analyzed (Participants) | 106
  Change from baseline in Borg score sitting at week 4 | 0.34 (1.94)
  Change from baseline in Borg score sitting at month 3: number analyzed (Participants) | 98
  Change from baseline in Borg score sitting at month 3 | 0.61 (2.08)
  Change from baseline in Borg score sitting month 6: number analyzed (Participants) | 46
  Change from baseline in Borg score sitting month 6 | 1.2 (1.87)
  Change from baseline in Borg score sitting at end of study: number analyzed (Participants) | 158
  Change from baseline in Borg score sitting at end of study | 1.07 (2.54)

9. Secondary Outcome: Number of Subjects Requiring Health and Home Care Resource Use
Description: The number of study subjects requiring Health and home care resource use was aggregated over the course of the study for each subject and summarised using descriptive statistics.
Time Frame: Baseline through study completion (2- 48 weeks after study entry)
Measure: Count of Participants; unit: Participants
Arm/Group | Levosimendan
Number analyzed (Participants) | 227
Participants | 95

10. Secondary Outcome: Subject's Status for Tracheostomy and Survival
Description: Number of patients with the need for tracheostomy or who died whilst on treatment from baseline to the end of the study was summarised using descriptive statistics.
Time Frame: Baseline to end of study (average 2-48 weeks after study entry
Population: Analysis was performed on the safety population which includes all subjects receiving at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Levosimendan
Number analyzed (Participants) | 227
Participants
  Number of participants who died from baseline to end of the study treatment | 5
  Number of participants requiring tracheostomy from baseline to the end of the study treatment | 0

11. Secondary Outcome: Health Care Service Use During the Study(Stays in Hospital)
Description: The number of night stays in hospital were recorded throughout the study using a diary given to the study subjects
Time Frame: From baseline to the end of the study(2-48 weeks after study entry)
Population: Analysis performed on the safety population defined as any subject receiving at least one dose of study treatment
Measure: Mean (Standard Deviation); unit: Nights
Arm/Group | Levosimendan
Number analyzed (Participants) | 227
Nights | 0.7 (2.7)

12. Secondary Outcome: Health Care Service Use During the Study(Visits to the Emergency Room)
Description: The number of visits to the emergency room were recorded throughout the study using a diary given to the study subjects
Time Frame: From baseline to the end of the study(2-48 weeks after study entry)
Population: Analysis performed on the safety population defined as any subject receiving at least one dose of study treatment
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Levosimendan
Number analyzed (Participants) | 227
visits | 0.1 (0.4)

13. Secondary Outcome: Health Care Service Use During the Study (Days Spent in an Institutional Facility)
Description: The number of days spent in an institutional facility were recorded throughout the study using a diary given to the study subjects
Time Frame: From baseline to the end of the study(2-48 weeks after study entry)
Population: Analysis performed on the safety population defined as any subject receiving at least one dose of study treatment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Levosimendan
Number analyzed (Participants) | 227
days | 4.7 (28.2)

ADVERSE EVENTS:
Time Frame: From signing informed consent until 14-25 days after the last study treatment administration, an average of 23.5 weeks.
Description: Four enrolled subjects did not start study treatment and are excluded from the safety population
Arm/Group | Levosimendan
All-Cause Mortality (participants affected / at risk) | 19/227
Serious Adverse Events (participants affected / at risk) | 44/227
Other Adverse Events (participants affected / at risk) | 215/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levosimendan (N=227)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysponea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 4 (5)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Cystitis bacterial (Infections and infestations) | 1 (1)
Systemic Viral Infection (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Lower Intestinal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Saliva altered (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Stoma Site Pain (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Subdural Hematoma (Injury, poisoning and procedural complications) | 1 (1)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1)
Meniscus Injury (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Euthanesia (General disorders) | 1 (1)
Back Pain (Metabolism and nutrition disorders) | 2 (2)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastasis to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal Mass (Renal and urinary disorders) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Oxygen Saturation decreased (Investigations) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levosimendan (N=227)
Fall (Injury, poisoning and procedural complications) | 25 (42)
Headache (Nervous system disorders) | 20 (28)
Tachycardia (Cardiac disorders) | 18 (20)
Dysponea (Respiratory, thoracic and mediastinal disorders) | 14 (15)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 13 (13)
Heart Rate Increased (Investigations) | 12 (12)
Dysphagia (Gastrointestinal disorders) | 11 (11)
Constipation (Gastrointestinal disorders) | 10 (11)
Nasopharyngitis (Infections and infestations) | 10 (11)
Diarrhoea (Gastrointestinal disorders) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Urinary Tract Infection (Infections and infestations) | 8 (9)
Oedema peripheral (General disorders) | 7 (8)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 6 (7)
Skin Laceration (Injury, poisoning and procedural complications) | 6 (7)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (7)
Insomnia (Psychiatric disorders) | 5 (5)
Anxiety (Psychiatric disorders) | 6 (6)
Dizziness (Nervous system disorders) | 6 (7)
Pyrexia (General disorders) | 5 (6)
Vomiting (Gastrointestinal disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/78/NCT03948178/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/78/NCT03948178/SAP_001.pdf